CLINICAL TRIAL: NCT01979770
Title: Association of Early Life Nutritional Related Exposures and Long-term Health and Cognitive Development Outcomes in Adolescents in Northeast, Thailand
Brief Title: Early Life Nutritional Exposures and Long-term Health and Cognitive Outcomes
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Tippawan Pongcharoen, Researcher, Mahidol University
Other Study IDs: MU-IRB2012/109.1611; COA 2013/008.1501 (Other: Mahidol University)
Record Dates: First submitted 2013-07-28; First posted 2013-11-08 (Estimated); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Overnutrition; Undernutrition
Keywords: Adolescent; Nutritional status; Body composition; Biochemical status
MeSH Terms: conditions — Overnutrition; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from blood specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adolescents: Adolescents who participated in an intervention trial of iron and zinc supplementation and a follow-up study at 9 years of age in 3 rural districts in Khon Kaen province, northeast of Thailand.

SUMMARY:
This study aims to investigate the relationship of the various exposures during infancy and childhood on later health and development of adolescents. Various exposures to be assessed include, but not limit to, nutritional status, body composition, energy expenditure, dietary intake, micronutrient status, breastfeeding, lifestyle, and other environment exposures.

The study will specifically aim to respond these research questions:

1.1 What are the factors associated with overweight, obesity, and stunted in adolescents? 1.2 What are the factors associated with increased risk of NCDs during adolescence? 1.3 What are the factors associated with cognitive functioning during adolescence? Since numerous variables were collected, additional research questions can be possibly studied or other interested variables can be included in the future.

DETAILED DESCRIPTION:
A longitudinal data were collected in children in the northeast of Thailand beginning at 4-6 months of age and every 2 months through 10-12 months of age while children had been given iron and/or zinc supplementation. Biochemical, anthropometric, socio-demographic, feeding practices, and maternal characteristics data were collected. Children were followed up at 9 years of age to assess the long-term consequences of supplementation and early life nutrition on cognitive functioning and growth. There is a need to continue the follow-up of this study in order to address the association between early nutritional exposures and risks of cardio-metabolic dysfunction and cognitive and behavioral development later in childhood, adolescence and adulthood. Thus, we propose to follow-up these children during adolescence to assess the relationship of early life nutrition and exposures during infancy and childhood and outcomes including nutritional status, cognitive functioning, and risk for non-communicable diseases (NCDs). Findings from this study could provide awareness and information in developing policies and timely interventions to maintain optimal nutritional status throughout vulnerable life stages and reduce risks of NCDs and disabilities later in life.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy children

Exclusion Criteria:

* none

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Adolescents who participated in an intervention trial of iron and zinc supplementation and a follow-up study at 9 years of age in 3 rural districts in Khon Kaen province, northeast of Thailand.
Sampling Method: Non-Probability Sample
Enrollment: 529 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-03-21 (Actual)

PRIMARY OUTCOMES:
Body composition | 1 year
  Body fat mass (kg), Body fat-free mass (kg) % body fat mass (%), % body fat-free mass (%)

SECONDARY OUTCOMES:
Cognition | 1 year
  IQ scores (IQ point)

OTHER OUTCOMES:
Cardio-vascular fitness | 1 year
  VO2max (L/min)

CONTACTS AND LOCATIONS:
Overall Officials: Tippawan Pongcharoen, Ph.D., Principal Investigator — Mahidol University
Locations (1):
- Institute of Nutrition, Mahidol University, Salaya, Changwat Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: Undecided